CLINICAL TRIAL: NCT03987841
Title: Intervention Mapping to Adapt a Mindfulness-based Intervention for Adults With Diabetes and Emotional Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Caroline Presley, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300003578; KL2TR003097 (NIH)
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Results first posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Type 2 Diabetes; Stress
Keywords: Diabetes distress; Mindfulness-based intervention; Diabetes self-management education
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrated MBSR/DSME intervention (Experimental): Integrated mindfulness-based stress reduction/diabetes self-management education intervention. Single-arm study, a group of participants meeting eligibility requirements will be invited to participate.
  Interventions: Behavioral: Integrated MBSR/DSME intervention

INTERVENTIONS:
Behavioral: Integrated MBSR/DSME intervention — Integrated mindfulness-based stress reduction/diabetes self-management education intervention. The intervention will comprise components of MBSR and DSME and will be delivered in a group setting with 8 weekly sessions. A trained masters-level interventionist will deliver the integrated intervention.

SUMMARY:
We will conduct a single-arm pilot study of an integrated mindfulness-based stress reduction (MBSR)/diabetes self-management education (DSME) intervention in a small group of participants, low-income adults with type 2 diabetes and diabetes distress. We will evaluate the preliminary efficacy, acceptability, and feasibility of the intervention.

DETAILED DESCRIPTION:
The intervention will comprise components of MBSR and DSME and will be delivered in a group setting with 8 weekly sessions. We anticipate enrollment of 30 participants, who will be adults with poorly controlled type 2 diabetes and elevated diabetes distress recruited from Cooper Green Mercy Health Systems, a safety-net health system serving residents of Jefferson County, Alabama. A trained masters-level interventionist will deliver the integrated intervention. The aim of the intervention is to reduce diabetes distress and improve glycemic control.

Participants will be assessed at baseline and 2 months. We will assess the preliminary efficacy of the intervention through pre/post evaluation of diabetes distress, diabetes self-management behaviors, and glycemic control as measured by hemoglobin A1c. Additionally, we will assess acceptability of the intervention through follow-up qualitative, focus groups with intervention participants; the feasibility of intervention delivery will be assessed using process measures.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Receipt of care at Cooper Green Mercy Healthcare System (CGMHS), one or more visits to primary care or diabetes clinic within the prior year
* An elevated point-of-care hemoglobin A1c (A1C) ≥7.5
* Presence of moderate diabetes distress (indicated by a score of ≥2 on the Diabetes Distress Scale)

Exclusion Criteria:

* Non-English speaking
* Currently pregnant
* Personal history or prior diagnosis of bipolar disorder, schizophrenia, or psychosis

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline A Presley, MD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Cooper Green Mercy Health Systems, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Integrated MBSR/DSME Intervention
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Integrated MBSR/DSME Intervention
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (6.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Diabetes Distress
Description: Measured by the diabetes distress scale (DDS), a 17-item self-report measure, assessing domains of emotional burden, physician-related distress, regimen-related distress, and interpersonal distress. The questionnaire will be administered to participants in English by a trained interviewer. The mean item score yields a possible score from 1 to 6; a score of <2 indicates little/no distress, 2 to 2.9 moderate distress, and ≥3 high distress.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrated MBSR/DSME Intervention
Number analyzed (Participants) | 5
score on a scale | 2.64 (0.94)

2. Primary Outcome: Diabetes Distress
Description: as for outcome 1
Time Frame: 2-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrated MBSR/DSME Intervention
Number analyzed (Participants) | 5
score on a scale | 2.19 (0.68)

3. Primary Outcome: Hemoglobin A1c (A1C)
Description: Participants will have a point-of-care A1C measured; A1C will be obtained by trained study personnel using finger-stick testing with the A1C Now+20 Test Kit (PTS diagnostics). A1C reports a % glycated hemoglobin level; a higher score indicates higher average blood glucose levels over the preceding 3 months. An A1C greater than or equal to 7.5% indicates poorly controlled type 2 diabetes.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Integrated MBSR/DSME Intervention
Number analyzed (Participants) | 5
percentage of glycosylated hemoglobin | 7.14 (0.88)

4. Primary Outcome: Hemoglobin A1c (A1C)
Description: Participants will have a point-of-care A1C measured; A1C will be obtained by trained study personnel using finger-stick testing with the A1C Now+20 Test Kit (PTS diagnostics). 1C reports a % glycated hemoglobin level; a higher score indicates higher average blood glucose levels over the preceding 3 months. An A1C greater than or equal to 7.5% indicates poorly controlled type 2 diabetes.
Time Frame: 2-months
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Integrated MBSR/DSME Intervention
Number analyzed (Participants) | 5
percentage of glycosylated hemoglobin | 7.24 (0.98)

5. Secondary Outcome: Diabetes Self-management Behaviors
Description: Measured by the Summary of Diabetes Self-Care Activities (SDSCA), a 10-item self-report measure that assesses diet (4-items), exercise (2-items), blood-glucose testing (2-items), and foot care (2-items). An example item is "How many of the last seven days have you followed a healthful eating plan?" Participants respond based on their self-care experience for the preceding week, from 0 to 7 indicating the number of days the participant performed the behavior. Each subscale is scored separately and scores are not combined. For each subscale, the score is the mean item score (i.e. mean number of days the activity was performed, range 0-7). A higher score indicates higher adherence to the self-care behavior. The questionnaire will be administered to participants in English by a trained interviewer.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Integrated MBSR/DSME Intervention
Number analyzed (Participants) | 5
units on a scale
  Diet | 3.96 (1.54)
  Exercise | 3.4 (2.36)
  Blood Glucose | 3.8 (2.41)
  Foot Care | 6.3 (1.57)

6. Secondary Outcome: Diabetes Self-management Behaviors
Description: as for outcome 5
Time Frame: 2-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Integrated MBSR/DSME Intervention
Number analyzed (Participants) | 5
units on a scale
  Diet | 4.4 (1.47)
  Exercise | 3.1 (1.82)
  Blood Glucose | 4.7 (2.20)
  Foot Care | 5.4 (2.50)

7. Secondary Outcome: Medication Adherence
Description: Participants will complete the Adherence to Refills and Medications - Diabetes (ARMS-D), an 11-item, self-report measure that includes medication-taking and refill subscales. Example item is "How often do you forget to take your diabetes medicine(s)?" Participants respond on a 4-point Likert scale from 1="none of the time" to 4="all of the time." Item responses are summed, combining subscales, yielding scores ranging from 11 to 44 (higher scores indicate greater difficulty with medication adherence). The questionnaire will be administered to participants in English by a trained interviewer.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrated MBSR/DSME Intervention
Number analyzed (Participants) | 5
score on a scale | 17 (9.54)

8. Secondary Outcome: Medication Adherence
Description: as for outcome 7
Time Frame: 2-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrated MBSR/DSME Intervention
Number analyzed (Participants) | 5
score on a scale | 16.2 (5.17)

9. Secondary Outcome: Acceptability of the Intervention to Participants: Semi-structured Interviews
Description: Acceptability will be assessed by conducting qualitative, semi-structured interviews with participants at the conclusion of the intervention. The interviews will gather participants' perspectives on the following: assessment of intervention content, perceived positive or negative effects, appropriateness of intervention duration and frequency, barriers to engagement, suggestions to improve the intervention, and overall satisfaction. Interviews will be recorded and transcribed. A combined inductive/deductive approach will be used for qualitative analysis, to identify themes reported by participants.
Time Frame: 2-months
Population: Not calculable value, based on qualitative analysis intervention acceptable to participants
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated MBSR/DSME Intervention
Number analyzed (Participants) | 5
Participants
  Handouts and study materials were easy to understand and useful for participants | 5
  Participants made changes related to mindful eating, physical activity, and managing stress | 5
  Participants reported main challenge was finding time to do activities outside of study sessions | 5
  Participant suggestion: more clearly linking discussions about stress and diabetes management | 5
  Participant suggestion: include more examples and opportunities to practice exercises | 5
  Participant suggestion: include multiple methods to access guidance for home practices | 5
  Overall satisfaction with program was high | 5

10. Secondary Outcome: Feasibility: Percentage of Screened Participants Who Are Eligible
Description: We will assess the percentage of screened participants who are eligible to participate in the study. Study staff will track the number of participants who are screened for participation and the number of participants who are eligible to participate.
Time Frame: Baseline
Population: This was total number of participants screened for eligibility.
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated MBSR/DSME Intervention
Number analyzed (Participants) | 16
Participants | 11

11. Secondary Outcome: Feasibility: Percentage of Eligible Participants Who Enroll
Description: We will assess the percentage of eligible participants who enroll in the study. Study staff will track the number of participants who are eligible for participation and the number of participants who enroll in the study.
Time Frame: Baseline
Population: This is the number of eligible participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated MBSR/DSME Intervention
Number analyzed (Participants) | 11
Participants | 5

12. Secondary Outcome: Feasibility: Distribution of Participants by Demographics
Description: We will collect demographics of study participants including age, race, ethnicity, and gender by participant self-report. This information will be obtained during a questionnaire administered to participants in English by a trained interviewer. We will use descriptive statistics to characterize the demographics of the study sample.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated MBSR/DSME Intervention
Number analyzed (Participants) | 5
Participants
  Non-Hispanic white male | 1
  Non-Hispanic Black female | 3
  Non-Hispanic Black male | 1

13. Secondary Outcome: Feasibility: Percentage of Sessions Attended
Description: We will track the number of sessions attended by each participant and calculate the percentage of overall sessions attended for each participant.
Time Frame: 2-months
Measure: Count of Participants; unit: Participants
Arm/Group | Integrated MBSR/DSME Intervention
Number analyzed (Participants) | 5
Participants
  100% attendance | 3
  85% attendance | 1
  71% attendance | 1

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Integrated MBSR/DSME Intervention
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
We experienced limitations in recruiting participants and delays in conducting the trial related to COVID (including interruptions in in-person care related to COVID). These factors resulted in smaller study sample than planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-10-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT03987841/Prot_SAP_ICF_000.pdf